CLINICAL TRIAL: NCT05013398
Title: Supporting the Mental Health Needs of Military Partners Through The Together Webinar Programme: Pilot Randomized Controlled Trial
Brief Title: The Together Webinar Programme For Military Partners
Acronym: TTP-Webinar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combat Stress (Other)
Collaborators: Royal British Legion (Unknown)
Responsible Party: Principal Investigator, Prof. Dominic Murphy, Head of research department, Combat Stress
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EGR17Q4\100016
Record Dates: First submitted 2021-07-29; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Psychological Distress
Keywords: Military partners; Mental Health Support; Online group-based support

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Together Webinar Programme (TTP-Webinar) (Experimental): Participants receive the six weekly session TTP-Webinar intervention.
  Interventions: Behavioral: The Together Webinar Programme
- Waitlist condition (No Intervention): Participants do not receive any intervention as part of waitlist condition. Note: Following the collection of measures at the follow-up time point, participants assigned to the waitlist condition were offered four TTP-Webinar groups to sign up to.

INTERVENTIONS:
Behavioral: The Together Webinar Programme — The TTP-Webinar consists of six hour-long sessions. Each session focuses on psychoeducation and self-management strategies for supporting veteran mental health difficulties as well as self-management tools to enhance partners' own wellbeing.
  The TTP-Webinar treatment protocol incorporates a range of techniques used in Cognitive Behavioral Therapy (CBT), Dialectical Behavioral Therapy (DBT), Compassion Focused Therapy (CFT), and Acceptance and Commitment Therapy (ACT).
  Other Names: TTP-Webinar
  Arms: The Together Webinar Programme (TTP-Webinar)

SUMMARY:
Military partners are at risk of mental health difficulties, including depression, anxiety and secondary traumatization. However, many partners face a range of barriers in accessing psychological support. As such, there remains a need to investigate how to make support for military partners more accessible.

The present study was a pilot randomized controlled trial (RCT) investigating the effectiveness of The Together Webinar Programme (TTP-Webinar) in reducing psychological distress and secondary trauma symptoms and improving quality of life among partners of veterans with PTSD and other mental health difficulties. The pilot RCT compared the TTP-Webinar intervention to a waitlist condition. The primary aim was to assess the acceptability and feasibility of offering web-based support to military partners and to investigate the efficacy of the remote-access support.

It was hypothesized that, compared to the waitlist condition, the TTP-Webinar would result in significant reductions in psychological distress and secondary symptoms, and improvements in overall quality of life.

DETAILED DESCRIPTION:
Evidence has found that living alongside a veteran suffering from mental health difficulties can have an adverse outcome on relationships and the health of family members. Military partners, in particular, have been highlighted as a high-risk group for developing mental health difficulties due to their close relationship with the veteran, exposure to adverse details of the veteran's military experiences and, in some cases, need to take on a caregiving role. Investigation of the impact on military partners suggests that they are an increased risk of depression, anxiety, alcohol use difficulties, as well as symptoms of secondary traumatization.

Despite an interest and need for mental health support among military partners, many face a range of barriers that prevent accessing and engaging in support. Such barriers include stigma around help seeking behaviors, difficulties in travelling to support venues, and work or childcare responsibilities that may limit their availability to engage with support. As such, there remains a need to make mental health support for military partners more accessible.

The Together Webinar Programme (TTP-Webinar) is a six-week online intervention developed to increase the accessibility of mental health support for military partners. TTP-Webinar was adapted from a five-week community-based TTP programme that was piloted across nine UK locations. Despite the community-based TTP programme demonstrating promising effects on mental health difficulties among military partners, the pilot revealed that many partners were unable to engage with support because of issues traveling to and from community centres around balancing other commitments.

The present study was a pilot randomized controlled trial (RCT) aimed at investigating the utility of TTP-Webinar as an online intervention to increase the accessibility of support. 60 partners of veterans with PTSD and other mental health difficulties were randomised to either the TTP-Webinar intervention (n = 30) or waitlist condition (n = 30). Measures of general psychological distress, secondary trauma symptoms and quality of life were administered at baseline, end of treatment, and one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Be over the age of 18
* Live in the UK
* Currently be in relationship with a veteran
* Provide written consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of the psychological distress on the General Health Questionnaire (GHQ-12) from baseline to end of treatment to 1-month follow-up | Baseline, end of treatment (6 weeks), and one-month follow-up.
  The GHQ-12 (Goldberg & Williams, 1988) is 12-item measure of symptoms of general psychological distress. Items are scoring using a 5-point Likert scale ranging from 0 ('Not at all'/'Much less than usual') to 4 ('Much more than usual'/'More so than usual'), indicating how much they have been bothered by symptoms within the past month. Six positive items are reverse scored, before calculating a total score with larger scores indicating greater psychological distress.
Change in symptoms of secondary traumatization on the Secondary Traumatic Stress Scale (STSS) from baseline to end of treatment to 1-month follow-up | Baseline, end of treatment (6 weeks), and one-month follow-up.
  The STSS (Bride et al., 2004) is a 17-item measure assessing symptoms of secondary traumatization. Items are scored on a 5-point Likert scale ranging from 0 ('Never') to 5 ('Very often'), indicating how much they have been bothered by symptoms within the past month. Total scores are created per subscales (avoidance, arousal, and intrusions) and across all subscales, with larger scores indicating greater secondary trauma symptoms.
Change in Quality of life (QoL) from baseline to end of treatment to 1-month follow-up. | Baseline, end of treatment (6 weeks), and one-month follow-up.
  QoL was assessed with a single item, using a scale ranging from 1 ('Very good') to 5 ('Very bad'). Scores were reverse scored, for larger scores to reflect greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Murphy, Principal Investigator — Combat Stress
Locations (1):
- Combat Stress, Leatherhead, Surrey, United Kingdom

REFERENCES:
- [Background] Thandi G, Oram S, Verey A, Greenberg N, Fear NT. Informal caregiving and intimate relationships: the experiences of spouses of UK military personnel. J R Army Med Corps. 2017 Aug;163(4):266-272. doi: 10.1136/jramc-2016-000679. Epub 2016 Dec 1. PMID 27909070
- [Background] Yambo T, Johnson M. An integrative review of the mental health of partners of veterans with combat-related posttraumatic stress disorder. J Am Psychiatr Nurses Assoc. 2014 Jan-Feb;20(1):31-41. doi: 10.1177/1078390313516998. Epub 2014 Jan 17. PMID 24441511
- [Background] Ray SL, Vanstone M. The impact of PTSD on veterans' family relationships: an interpretative phenomenological inquiry. Int J Nurs Stud. 2009 Jun;46(6):838-47. doi: 10.1016/j.ijnurstu.2009.01.002. Epub 2009 Feb 7. PMID 19201406
- [Background] Sayers SL, Farrow VA, Ross J, Oslin DW. Family problems among recently returned military veterans referred for a mental health evaluation. J Clin Psychiatry. 2009 Feb;70(2):163-70. doi: 10.4088/jcp.07m03863. Epub 2009 Feb 10. PMID 19210950
- [Background] Murphy D, Palmer E, Busuttil W. Mental Health Difficulties and Help-Seeking Beliefs within a Sample of Female Partners of UK Veterans Diagnosed with Post-Traumatic Stress Disorder. J Clin Med. 2016 Aug 1;5(8):68. doi: 10.3390/jcm5080068. PMID 27490576
- [Background] Murphy D, Spencer-Harper L, Turgoose D. Exploring the feasibility of supporting UK partners living alongside veterans with PTSD: A pilot study of the Together Programme (TTP). Journal of Family Medicine. 2019; 1(2): 30-41.
- [Derived] Hendrikx LJ, Murphy D. Supporting the Mental Health Needs of Military Partners Through the Together Webinar Program: Pilot Randomized Controlled Trial. JMIR Ment Health. 2021 Oct 12;8(10):e25622. doi: 10.2196/25622. PMID 34636734